CLINICAL TRIAL: NCT00003289
Title: A Phase I and Pharmacologic Study of UCN-01 (NSC638850)
Brief Title: UCN-01 in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: JHOC-J9814, CDR0000066221; U01CA070095 (NIH); P30CA006973 (NIH); JHOC-98012305; NCI-T97-0083
Record Dates: First submitted 1999-11-01; First posted 2004-05-21 (Estimated); Last update posted 2010-08-09 (Estimated); Status verified 2010-08

CONDITIONS: Leukemia; Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: Waldenstrom macroglobulinemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia; unspecified adult solid tumor, protocol specific; refractory hairy cell leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; prolymphocytic leukemia; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Leukemia, Prolymphocytic; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — 7-hydroxystaurosporine

INTERVENTIONS:
Drug: 7-hydroxystaurosporine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of UCN-01 in treating patients with advanced cancer that has not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity profile, dose limiting toxicity, and maximum tolerated dose of UCN-01 administered as a 3, 2, or 1 hour infusion every 4 weeks for patients with advanced solid tumor malignancies and chronic lymphoproliferative disorders. II. Investigate the pharmacokinetics and cellular pharmacodynamics of UCN-01 administered on this schedule in these patients. III. Obtain preliminary evidence of the antitumor activity of UCN-01 in this patient population.

OUTLINE: This is dose escalation study. Patients receive UCN-01 by intravenous infusions over 3, 2 or 1 hour(s) every 4 weeks. The first dose level is administered over 3 hours, the next dose level is administered over 2 hours, and the next and subsequent dose levels are administered over 1 hour. One patient is treated at each dose level until unacceptable toxicity is observed. An additional 2 patients are then entered at that dose level. If dose limiting toxicity (DLT) is experienced in 1 of 3 patients, 3 additional patients are accrued at that dose level. If 2 or more patients experience DLT, the maximum tolerated dose has been surpassed and a total of 6 patients must be treated at the previous dose level. If no patients develop DLT, the dose is escalated in successive cohorts of 3 patients per dose level. Patients are followed for 4 weeks after each drug administration before subsequent patients can be entered at the next higher dose level. Patients are followed for 2 months after their last dose of UCN-01.

PROJECTED ACCRUAL: Approximately 36 patients will be accrued into this study over 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed malignancy that is refractory to standard therapy or for which no standard therapy exists Low grade lymphoproliferative disorder defined as: Chronic lymphocytic leukemia/small lymphocytic lymphoma Waldenstrom's macroglobulinemia Follicular lymphoma (small cleaved, mixed, and large cell) Mantle cell lymphoma Prolymphocytic leukemia (T and B type) Cutaneous T cell non-Hodgkin's lymphoma Marginal zone lymphoma and variants Hairy cell leukemia variants MALT lymphomas Patients with low grade lymphoproliferative disorders must have received at least 1 or more treatment regimens and must not be eligible for potentially curative treatments (i.e., bone marrow transplantation) No HTLV-1 associated lymphomas, Burkitt's or small non-cleaved lymphomas, transplant related lymphoproliferative disorders, Hodgkin's disease, diffuse large cell lymphoma, or multiple myeloma No primary brain tumors or history of brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count greater than 1,500/mm3 Platelet count greater than 100,000/mm3 Hemoglobin at least 8.0 g/dL Hepatic: Bilirubin no greater than 1.2 mg/dL AST/ALT less than 2.5 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: No history of unstable or newly diagnosed angina pectoris No myocardial infarction within the last 6 months No New York Heart Association class II-IV congestive heart failure Neurologic: No grade 2 or greater peripheral neuropathy Pulmonary: No grade 2 or greater pulmonary toxicity (dyspnea on significant exertion) Other: HIV negative No autoimmune hemolytic anemia Must be able to have a central venous access catheter No active infections requiring oral or intravenous antibiotics No medical or psychiatric problems unrelated to the malignancy that may limit compliance with study, expose patient to undue risk, or confound toxicity assessment Not pregnant or nursing Adequate contraception is required of all fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 1 month since prior platelet or red blood cell transfusions Chemotherapy: At least 6 weeks since nitrosoureas or mitomycin At least 4 weeks since other chemotherapy No investigational or standard chemotherapy for at least 2 months after completion of last dose of UCN-01 Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since radiotherapy Surgery: At least 4 weeks since major surgery Other: No concurrent anticonvulsant medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-06

CONTACTS AND LOCATIONS:
Overall Officials: Ross C. Donehower, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Johns Hopkins Oncology Center, Baltimore, Maryland, United States